CLINICAL TRIAL: NCT00895323
Title: Phase I Study of Preoperative Detection of Colorectal Carcinoma With Bispecific Antibody Pretargeting
Brief Title: Bispecific Antibody in Finding Tumor Cells in Patients With Colorectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Garden State Cancer Center at the Center for Molecular Medicine and Immunology (Other)
Responsible Party: Sylvia Gargiulo, Garden State Cancer Center and Center for Molecular Medicine and Immunology
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000636332; CMMI-C-071A-07
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-07

CONDITIONS: Colorectal Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Enzyme-Linked Immunosorbent Assay

INTERVENTIONS:
Other: enzyme-linked immunosorbent assay
Other: pharmacological study
Procedure: whole-body scintigraphy
Radiation: iodine I 131-labeled anti-CEA/anti-HSG bispecific monoclonal antibody TF2

SUMMARY:
RATIONALE: Diagnostic procedures, such as radionuclide imaging using bispecific antibody, may help find colorectal cancer cells and learn the extent of disease.

PURPOSE: This phase I trial is studying how well a bispecific antibody works in finding tumor cells in patients with colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the pharmacokinetics and tissue distribution of anti-CEA x anti-HSG bispecific monoclonal antibody TF2 in patients with colorectal cancer.

OUTLINE: This is a multicenter study.

Patients receive iodine I 131-labeled anti-CEA x anti-HSG bispecific monoclonal antibody TF2 (^131I-TF2) IV over 10-20 minutes on day 1. Patients also undergo whole-body external scintigraphy at various times during the study.

Blood samples are collected at baseline and periodically after ^131I-TF2 infusion for pharmacokinetic studies and ^131I-TF2 biodistribution by ELISA and radioactivity measurements.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer

  * Radiological documentation of disease is preferred, but not required

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Life expectancy ≥ 3 months
* WBC ≥ 3,000/mm³
* Neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Serum creatinine normal
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST/ALT < 2 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 1 month after completion of study therapy
* No medical conditions that might prevent full participation in protocol-required testing or follow-up
* No institutionalized patients (e.g., in prisons or mental health institutions)

PRIOR CONCURRENT THERAPY:

* No concurrent chemotherapy or treatments that would compromise the safety and efficacy of protocol assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics
Tissue distribution

CONTACTS AND LOCATIONS:
Overall Officials: Aiwu R. He, MD, Principal Investigator — Lombardi Comprehensive Cancer Center
Locations (1):
- Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia, United States